CLINICAL TRIAL: NCT04518501
Title: Fuzuloparib Plus Arsenic Trioxide in Patients With Platinum Resistance Relapsed Ovarian Cancer
Brief Title: Fuzuloparib Arsenic Trioxide Platinum Resistance Relapsed Ovarian Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Xing Xie (Other)
Responsible Party: Sponsor-Investigator, Xing Xie, profressor, Women's Hospital School Of Medicine Zhejiang University
Organization: Women's Hospital School Of Medicine Zhejiang University (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CESM023
Record Dates: First submitted 2020-08-16; First posted 2020-08-19 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Efficacy and Safety
Keywords: PARPI; Arsenic Trioxide; High Grade Serous Carcinoma; High Grade Endometria Carcinoma; Platinum-resistant Ovarian Cancer; Fuzuloparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- study group (Experimental): Fuzuloparib Capsules plus table Arsenic Trioxide po
  Interventions: Drug: Arsenic trioxide Tablet +Fuzuloparib Capsules

INTERVENTIONS:
Drug: Arsenic trioxide Tablet +Fuzuloparib Capsules — Arsenic trioxide Tablet : 0.27*9 tid po consecutive 21 days with 1 week rest． Fuzuloparib Capsules: 150 mg bid po

SUMMARY:
Ovarian cancer is the leading cause of death from gynecologic tumors in the western world. Most patients have relapses, and responses to subsequent therapies are generally short-lived. Currently, the population that can benefit from PARPi is mainly focusing on BRCAm, then homologous-recombination deficiency patients. Limited data revealed the ORR was only 3-4% in homologous recombination proficiency patients with PARPi therapy. New treatments are urgently needed to improve patient outcomes.

To explore the efficacy and safety of Fuzuloparib in combination with Arsenic trioxide therapy in platinum-resistance relapsed Ovarian cancer patients.

DETAILED DESCRIPTION:
Ovarian cancer is the leading cause of death from gynecologic tumors in the western world. Most patients have relapses, and responses to subsequent therapies are generally short-lived. Currently, the population that can benefit from PARPi is mainly focusing on BRCAm, then homologous-recombination deficiency patients. Limited data revealed the ORR was only 3-4% in homologous recombination proficiency patients with PARPi therapy. New treatments are urgently needed to improve patient outcomes.

The investigators' studies have shown that combination therapy with Fuzuloparib and Arsenic trioxide demonstrated a synergistic anti-tumor effect in BRCAness/HR-proficiency ovarian cancer cells:

Firstly, CCK8 and clone formation assays showed that the combination of Fuzuloparib and Arsenic trioxide produced notable tumor cell growth inhibition than either single agent in SKOV3 and CAOV3 cells.

Further, the combination therapy resulted in significantly increased level of γ-H2AX and decreased level of RAD51 by IF.The investigators also found that combination therapy could remarkably induced cell apoptosis, which is associated with induction of cleave-PARP and reduction of p-AKT, when compared with either single drug. (Data not published) Therefore, the investigators hypothesis is that for those platinum-resistance relapsed patients who have received at least twice platinum-based chemotherapy, patients with combinate therapy will get 25% of ORR. And platinum-resistance in combination with Arsenic trioxide therapy is well tolerated.

ELIGIBILITY:
Inclusion Criteria:

* 18-70years old;
* High grade (serous or endometrioid) epithelial ovarian cancers, fallopian tube or primary peritoneal carcinoma;
* Patients received at least two lines of platinum-containing chemotherapy, with recurrence occurring within six months after the last chemotherapy dose, or were platinum-refractory patients who have undergone at least two cycles of platinum-based chemotherapy;
* Measurable disease as per RECIST 1.1
* ECOG 0-2;
* Life expectancy ≥12 weeks;
* Confirmation of BRCA1/2 mutation status;
* PARPi naive;
* LVEF ≥ 50%;
* Bone Marrow Function: ANC：≥1.5×109/L； PLT：≥100×109/L；Hb: ≥90g/L;
* Liver and renal function:Serum creatinine ≤ normal upper limit (ULN) 1.5times; aspartate aminotransferase (AST) and alanine aminotransferase (ALT)≤ULN 2.5times, or <ULN 5times in the presence of liver metastasis; total bilirubin (TBil) level≤ ULN 1.5 times, or ≤ ULN 2.5times if Gilbert's syndrome are present;
* The childbearing age subjects must agree to take effective contraceptive measures during the trial; the serum or urine pregnancy test must be negative, non-lactating;
* Signed the informed consent;

Exclusion Criteria:

* Prior treatment with PARP inhibitors except under specific conditions: 1. Patients who previously received PARP inhibitor (PARPi) therapy without disease progression during treatment, but discontinued due to reasons such as treatment cost or adherence issues; 2. Patients who received only one prior PARPi therapy (excluding fuzuloparib), with maintenance therapy lasting ≥ 12 months. In both cases, the time since the last PARPi treatment must be >6 months prior to study enrollment;
* Patients who had previously received >20% bone marrow radiotherapy in 1 week;
* Other malignant tumors have been found in the past 5 years,except for cured cervical carcinoma in situ, non melanoma of the skin;
* Uncontrolled systemic infection requiring anti-infective treatment;
* Allergies to the Fuzuloparib or Arsenic Trioxide or their excipients or intolerant patients;
* Subjects with ≥2 grade peripheral neuropathy according to CTCAE V 4.03;
* Researchers think it is not suitable for enrolling.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2024-12-03 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
ORR | From date of randomization until PD or death from any cause, assessed up to 36 months.
  ORR is defined as the rate of CR or PR, as determined by IRC using RECIST v1.1 criteria among patients with at least one target lesion. Activity was also described in women with nontarget lesions only and in women without any tumor lesion but with elevated CA-125 levels before starting treatment.

SECONDARY OUTCOMES:
OS | From date of randomization until the date of death from any cause, or date of last follow-up for patients still alive, assessed up to 36 months]
  overall survival
PFS | From date of randomization until the date of first documented progression or death from any cause, whichever occurred first, or last follow-up for patients alive without progression, assessed up to approximately 36 months
  PFS is defined as the time from randomization to the first occurrence of PD, as determined by the investigator using RECIST v1.1, or death from any cause during the study, whichever occurs first.
the incidence and severity of adverse reactions | A summary of adverse events of each cycle,from date of administration of drugs until 30 days after the last chemotherapy or progression,whichever came first,assessed up to 36 months
  Evaluate the adverse reactions rate of drugs assessed by number and severity of adverse events in the treatment.
quality of life assessment | It will be assessed at baseline and before the administration of drugs at each first day of every two chemotherapy cycles, up to 6 cycles,each cycle is 28days.
  according to the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire C30 (QLQ-C30).The basic content of life quality assessment includes: physical health, mental health, social function, disease status and overall health perception.

CONTACTS AND LOCATIONS:
Locations (1):
- Women's Hospital School Of Medicine Zhejiang University, Zhejiang, Hangzhou, China